CLINICAL TRIAL: NCT00382681
Title: Clinical Evaluation of the Safety and Efficacy of an Investigational Multi-Purpose Disinfecting Solution Compared to a Marketed Multi-Purpose Solution for Care of Soft Contact Lenses
Brief Title: Evaluation of an Investigational Multi-Purpose Disinfecting Solution for Care of Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-03-41
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Contact Lens Care
Keywords: Contact Lens Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FID 107027 (Experimental): Contact lens solution used as instructed for 90 days.
  Interventions: Device: FID 107027 Multi-Purpose Disinfecting Solution
- ReNu MultiPlus (Active Comparator): Contact lens solution used as instructed for 90 days.
  Interventions: Device: ReNu MultiPlus Multi-Purpose Solution No Rub Formula

INTERVENTIONS:
Device: FID 107027 Multi-Purpose Disinfecting Solution — Investigational, multi-purpose disinfecting solution intended for use in cleaning, rinsing, conditioning, disinfecting, and storing soft contact lenses.
  Arms: FID 107027
Device: ReNu MultiPlus Multi-Purpose Solution No Rub Formula — Commercially marketed product indicated for cleaning, rinsing, disinfecting, and storing soft contact lenses.
  Arms: ReNu MultiPlus

SUMMARY:
The objective of the study was to clinically evaluate the safety and effectiveness of a new multi-purpose disinfecting solution for soft contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Successful daily wear of FDA Group I or IV lenses on a two-week or longer replacement schedule for at least one month.
* Use of a multi-purpose solution only as the pre-study care regimen for at least one month (rewetting drops use is also acceptable).
* Successful lens wear for at least 8 hours per day.
* Vision correctable to 20/30.
* Normal eyes - no current ocular abnormalities that prevent successful contact lens wear.
* No corneal surgery within the past 12 months.
* No systemic disease that affects that eye or that could be worsened by the use of contact lenses or solutions.
* No over-the-counter or prescription ocular medication.
* No enrollment in another clinical study within 30 days prior to enrollment.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2004-07; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Lens Cleanliness - Residual lens lysozyme (HPLC) at Day 90 on Group IV lenses | Day 90

SECONDARY OUTCOMES:
Average Lens Wearing Time | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Napier, Study Director — Alcon Research
Locations (1):
- Elkin, Elkin, North Carolina, United States